CLINICAL TRIAL: NCT01186341
Title: BraveNet Multi-Center Study on Integrative Medicine Treatment Approaches for Pain
Acronym: SIMTAP
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: The Bravewell Collaborative (Other); Alliance Institute for Integrative Medicine (Other); Allina Health System (Other); University of Maryland (Other); Beth Israel Medical Center (Other); Thomas Jefferson University (Other); University of California, San Francisco (Other); Scripps Clinic (Other); Venice Family Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00018346
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2011-06

CONDITIONS: Chronic Pain
Keywords: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Pain: New or existing patients of the center who are seeking their initial treatment at the Integrative Medicine center for chronic pain (chronic > 3 months) who report their average pain level over the past month to be at least a 4 of 10 on the Visual Analog Scale.

SUMMARY:
Preliminary results from an ongoing cross-sectional survey of nine of the BraveNet Outpatient Clinics indicate that pain was the leading reason for patient visits. As a precursor to a large multi-site clinical trial, this study aims to determine the feasibility of collecting outcomes data on integrative treatment for pain. These preliminary data will also provide an estimation of effect size for powering the multi-site clinical trial.

DETAILED DESCRIPTION:
Integrative medicine (IM) provides a comprehensive approach to care in which healing and wellness of the whole person are the foremost goals. IM is not simply complementary and alternative medicine (CAM), but it stresses patient-centered, healing-oriented care that emphasizes the patient-caregiver relationship.

Little is known about the health outcomes of patients who present to an IM center and undergo a variety of treatment modalities to treat a specific condition. Adequately capturing and describing IM patient outcomes is a challenge for many reasons. First, given the whole person focus of IM, multiple domains of outcomes must be considered including physical, psychological, social, and spiritual. Second, since the patient-centric notion of individualized care is seminal to IM, IM outcomes must allow for patient-reported outcomes. Finally, the complexity of whole system care creates a natural barrier when measuring IM efficacy. Whole systems of care theoretically rely on synergistic and inseparable components and conceptualize the patient-practitioner interaction as a key component of care.

The Bravewell Integrative Medicine Research Network (BraveNet) is a practice-based research network of nine leading integrative medicine centers around the U.S. collaborating in clinical outcomes research to increase the knowledge and evidence-base of IM. These centers may differ in terms of patient population, medical conditions seen, IM services offered, and treatment outcomes, but all are committed to the provision of integrative care.

Preliminary results from an ongoing cross-sectional survey of nine of the BraveNet Outpatient Clinics indicate that pain was the leading reason for patient visits. As a precursor to a large multi-site clinical trial, this study aims to determine the feasibility of collecting outcomes data on integrative treatment for pain. These preliminary data will also provide an estimation of effect size for powering the multi-site clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be men and women aged 18 and over.
* Patient Status: Participants are eligible if they are new or existing patients of the center who are seeking their initial treatment at the Integrative Medicine center for chronic pain (chronic > 3 months) who report their average pain level over the past month to be at least a 4 of 10 on the VAS.
* English or Spanish Literacy: Ability to read and write English or Spanish as confirmed by the site personnel and ability to provide informed consent.
* Subject must provide written informed consent before initiation of any study-related procedures.
* Subject must be able to understand and comply with the requirements of the study, as judged by the investigator.

Exclusion Criteria:

* A subject will not be eligible if he/she is unable to provide Informed Consent.
* Inability to read and write in English or Spanish.
* Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the Investigator, unacceptably increase the patients risk by participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending one of the nine Integrative Medicine Clinics of the BraveNet research network.
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of assessing the impact of IM intervention on chronic pain | 24 weeks
  As measured by the number of patients approached to participate, number who refuse to participate, reasons for refusal, and the number of people who provide consent.

SECONDARY OUTCOMES:
Quality of Life | 24 weeks
  As measured by self report on a questionnaire
Sense of control | 24 weeks
  As measured by a Visual Analog Scale
Depression and Stress | 24 weeks
  As measured by self report questionnaires such as the depression (The Center for Epidemiologic Studies Depression Scale (CES-D)and stress (The Perceived Stress Scale - 4)
Inflammatory Marker and Vitamin D | 24 weeks
  High-sensitivity C reactive protein (hs-CRP) and 25-hydroxy-vitamin D levels at baseline and 12 weeks
Health services utilization | 24 weeks
  As measured by self report of health services(including medications and supplements).
Work productivity and activity impairment | 24 weeks
  As measured by the Work Productivity and Activity Impairment (WPAI) survey.
Estimate the effect size of IM interventions for reducing pain in chronic pain patients | 24 weeks
  As measured by the Pain-Visual analog scale of average and worst pain and (total) Brief Pain Inventory (BPI) interference scale

CONTACTS AND LOCATIONS:
Overall Officials: Rowena Dolor, MD, Principal Investigator — Duke Clinical Research Institute; Ruth Wolever, PhD, Principal Investigator — Duke Integrative Medicine Center
Locations (9):
- United States (9):
  - Scripps Center for Integrative Medicine, La Jolla, California
  - UCSF Osher Center for Integrative Medicine, San Francisco, California
  - Venice Family Clinic Simms/Mann Health and Wellness Center, Santa Monica, California
  - University of Maryland Center for Integrative Medicine, Baltimore, Maryland
  - Penny George Institute for Health and Healing, Minneapolis, Minnesota
  - The Continuum Center for Health and Healing, New York, New York
  - Duke Integrative Medicine, Durham, North Carolina
  - Alliance Center for Integrative Medicine, Cincinnati, Ohio
  - Jefferson-Myrna Brind Center of Integrative Medicine, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Abrams DI, Dolor R, Roberts R, Pechura C, Dusek J, Amoils S, Amoils S, Barrows K, Edman JS, Frye J, Guarneri E, Kligler B, Monti D, Spar M, Wolever RQ. The BraveNet prospective observational study on integrative medicine treatment approaches for pain. BMC Complement Altern Med. 2013 Jun 24;13:146. doi: 10.1186/1472-6882-13-146. PMID 23800144